CLINICAL TRIAL: NCT02395627
Title: Reversing Therapy Resistance With Epigenetic-immune Modification: Phase II Trial of Vorinostat, Tamoxifen and Pembrolizumab in Hormone Receptor Expressing Advanced Breast Cancer
Brief Title: Reversing Therapy Resistance With Epigenetic-Immune Modification
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient efficacy in an unselected patient population
Sponsor: University of California, San Francisco (Other)
Collaborators: Avon Foundation (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 147523; NCI-2015-00815 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2015-03-17; First posted 2015-03-23 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Breast Neoplasms
Keywords: Hormone Therapy Resistant; Estrogen Receptor-Positive; Estrogen Receptor-Negative
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; Vorinostat; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pembrolizumab Cycle 1 (Group A) (Experimental): Tamoxifen: 20 mg daily orally (starting at Cycle 1) Vorinostat: 400 mg 5 days every 7 orally (starting at Cycle 1) Pembrolizumab: 200 mg every 3 weeks intravenously (starting at Cycle 1)
  Interventions: Drug: Tamoxifen; Drug: Vorinostat; Drug: Pembrolizumab
- Pembrolizumab Cycle 2 (Group B) (Experimental): Tamoxifen: 20 mg daily orally (starting at Cycle 1) Vorinostat: 400 mg 5 days every 7 orally (starting at Cycle 1) Pembrolizumab: 200 mg every 3 weeks intravenously (starting at Cycle 2)
  Interventions: Drug: Tamoxifen; Drug: Vorinostat; Drug: Pembrolizumab
- Pembrolizumab Cycle 1 (Group C) (Experimental): Vorinostat: 400 mg 5 days every 7 orally (starting at Cycle 1) Pembrolizumab: 200 mg every 3 weeks intravenously (starting at Cycle 1)
  Interventions: Drug: Vorinostat; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Tamoxifen
  Other Names: Nolvadex
  Arms: Pembrolizumab Cycle 1 (Group A); Pembrolizumab Cycle 2 (Group B)
Drug: Vorinostat
  Other Names: Zolinza
Drug: Pembrolizumab
  Other Names: Keytruda

SUMMARY:
The investigators propose a randomized two arm trial, using Simon's 2-stage design, in ER+ patients with therapy resistant breast cancer to test the optimal sequence and dosing of epigenetic immune priming in hormone therapy resistance breast cancer. A third arm (Arm C) will include ER-negative patients who will follow the concurrent priming, but exclude tamoxifen. The two arms all include vorinostat, tamoxifen, and pembrolizumab to evaluate

* Sequential priming - begin pembrolizumab in Cycle 1 (Arm B and Arm C) and,
* Concurrent priming with maximal dosing of both epigenetic and immune modulators- begin pembrolizumab on day 1 in Cycle 2 (Arm A)

DETAILED DESCRIPTION:
Unique aspects of this study:

This is the first study to look at the response of hormone therapy resistance breast cancer to epigenetic immune priming. It is also the first study to look at the combination of an Histone deacetylase (HDAC) inhibitor (vorinostat), an anti-estrogen (tamoxifen) and a PD-1 inhibitor, pembrolizumab in pre or postmenopausal patients with ER+ advanced breast cancer with progression on multiple prior therapies.

Recent preclinical studies have further suggested that epigenetic priming may be even more effective in ER-negative tumors that do not respond to immune check point inhibitors or have low PD-1/PD-L1 expression. The goal of this study is to demonstrate that Vorinostat can increase PD-1 and PD-L1 expression.

In a third arm the study will evaluate the role of epigenetic priming in tumors that are ER-negative.

ELIGIBILITY:
Inclusion Criteria:

* Pre and postmenopausal women or men with stage IV ER+ breast cancer histological or cytological confirmation

ER-positive tumors

* Progressed after at least one line of hormonal therapy
* Any number of prior chemotherapy in the metastatic setting
* Any number of prior hormonal therapies.
* human epidermal growth factor receptor 2 (HER2) positive or negative

ER-Negative tumors

* PD-L1 low, high or unknown
* Progression after prior PD-1 or PD-L1 inhibitors allowed
* HER2 positive or negative
* 18 years or older
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2.
* Understand and voluntarily sign an informed consent prior to any study-related assessments or procedures are conducted and are able adhere to the study visit schedule and other protocol requirements.
* Consent to paired tumor biopsy, for accessible tumors
* Measureable tumor by RECIST criteria v.1.1
* Archived tumor tissue (minimum of 8 slides for paraffin-embedded tumor tissue) for assessment of tumor-based biomarkers and immune score is required for eligibility.
* Per Good Clinical Practice, any toxicity related to prior therapies that, in the opinion of the investigator, would potentially be worsened with anti-PD1 therapy should be resolved to less than Grade 1
* Adequate organ function within 14 days of study start:
* Absolute neutrophil count (ANC) ≥ 1.5 X 109/L
* Hemoglobin (Hgb) ≥9g/dL (may transfuse if clinically indicated)
* Platelets (plt) ≥ 100 x 109/L
* Potassium within normal range, or correctable with supplements;
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x Upper Limit Normal (ULN) or ≤5.0 x ULN if liver tumor is present;
* Serum total bilirubin ≤ 1.5 x ULN
* Serum creatinine ≤ 1.5 x ULN, or 24-hr clearance ≥ 60ml/min; and
* Females of child-bearing potential (defined as a sexually mature women who):
* Has not undergone a hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or,
* Has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time during the preceding 24 consecutive months).
* Must have negative serum pregnancy test within 7 days before starting study treatment in females of childbearing potential (FCBP) and willingness to adhere to acceptable forms or birth control (a physician- approved contraceptive method (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner).
* Male subjects with female partner of childbearing potential must agree to the use of a physician-approved contraceptive method throughout the course of the study

Exclusion Criteria:

* Any significant medical condition, laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
* Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
* Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Patients may continue on ovarian suppression
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Any condition that confounds the ability to interpret data from the study.
* Symptomatic central nervous system metastases. Subjects with brain metastases that have been previously treated and are stable for 6 weeks are allowed.
* Persistent diarrhea or malabsorption ≥ NCI CTCAE grade 2, despite medical management.
* Unstable angina, significant cardiac arrhythmia, or New York Heart Association (NYHA) class 3 or 4 congestive heart failure.
* Prior systemic cancer-directed treatments or investigational modalities ≤ 5 half-lives or 4 weeks, whichever is shorter, prior to starting study drug or who have not recovered from side effects of such therapy (except alopecia).
* Has an active auto-immune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Active and ongoing steroid use, except for non-systemically absorbed treatments (such as inhaled or topical steroid therapy for asthma, Chronic Obstructive Pulmonary Disease (COPD), allergic rhinitis).
* Major surgery ≤ 2 weeks prior to starting a study drug or who have not recovered from side effects of such therapy.
* Pregnant or breast feeding.
* Known Human Immunodeficiency Virus (HIV) infection and/or Hepatitis B or C positive.
* Known hypersensitivity to pembrolizumab or any of its excipients.
* Has received a live vaccine within 30 days prior to the first dose of trial treatment.
* Patients receiving medications or substances that are strong inhibitors or inducers of CYP450 enzyme(s) are ineligible.
* Pregnant women are excluded from this study because vorinostat, tamoxifen and PD-1 are drug classes with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother, breastfeeding should be discontinued if the mother is treated with vorinostat, tamoxifen and PD-1 inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-05-04 (Actual); Primary Completion 2019-06-08 (Actual); Study Completion 2019-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Munster, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco Medical Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Terranova-Barberio M, Pawlowska N, Dhawan M, Moasser M, Chien AJ, Melisko ME, Rugo H, Rahimi R, Deal T, Daud A, Rosenblum MD, Thomas S, Munster PN. Exhausted T cell signature predicts immunotherapy response in ER-positive breast cancer. Nat Commun. 2020 Jul 17;11(1):3584. doi: 10.1038/s41467-020-17414-y. PMID 32681091

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab Cycle 1 (Group A): Tamoxifen: 20 mg daily orally (starting at Cycle 1) Vorinostat: 400 mg 5 days every 7 orally (starting at Cycle 1) Pembrolizumab: 200 mg every 3 weeks intravenously (starting at Cycle 1)
  Tamoxifen
  Vorinostat
  Pembrolizumab
- Pembrolizumab Cycle 2 (Group B): Tamoxifen: 20 mg daily orally (starting at Cycle 1) Vorinostat: 400 mg 5 days every 7 orally (starting at Cycle 1) Pembrolizumab: 200 mg every 3 weeks intravenously (starting at Cycle 2)
  Tamoxifen
  Vorinostat
  Pembrolizumab
- Pembrolizumab Cycle 1 (Group C): Vorinostat: 400 mg 5 days every 7 orally (starting at Cycle 1) Pembrolizumab: 200 mg every 3 weeks intravenously (starting at Cycle 1)
  Vorinostat
  Pembrolizumab
Period: Overall Study
Arm/Group | Pembrolizumab Cycle 1 (Group A) | Pembrolizumab Cycle 2 (Group B) | Pembrolizumab Cycle 1 (Group C)
Started | 18 | 16 | 4
Completed | 15 | 13 | 4
Not Completed | 3 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0
Not completed — Did not receive pembrolizumab | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pembrolizumab Group A: Estrogen Receptor Positive (ER+) participants
  Tamoxifen: 20 mg daily orally (starting at Cycle 1) Vorinostat: 400 mg 5 days every 7 orally (starting at Cycle 1)
  Group A Pembrolizumab: 200 mg every 3 weeks intravenously (starting at Cycle 1)
- Pembrolizumab Group B: Estrogen Receptor Positive (ER+) participants
  Tamoxifen: 20 mg daily orally (starting at Cycle 1) Vorinostat: 400 mg 5 days every 7 orally (starting at Cycle 1)
  Group B Pembrolizumab: 200 mg every 3 weeks intravenously (starting at Cycle 2)
- Pembrolizumab Group C: Estrogen Receptor Negative (ER-) participants
  Vorinostat: 400 mg 5 days every 7 orally (starting at Cycle 1) Pembrolizumab: 200 mg every 3 weeks intravenously (starting at Cycle 1)
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab Group A | Pembrolizumab Group B | Pembrolizumab Group C | Total
Number analyzed (Participants) | 18 | 16 | 4 | 38
Age, Customized [Count of Participants; unit: Participants]
  30-39 years old | 2 | 4 | 0 | 6
  40-49 years old | 4 | 3 | 1 | 8
  50-59 years old | 5 | 3 | 2 | 10
  60-69 years old | 4 | 5 | 1 | 10
  70-79 years old | 2 | 1 | 0 | 3
  80-89 years old | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 15 | 4 | 37
  Male | 0 | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 14 | 13 | 2 | 29
  Unknown or Not Reported | 3 | 3 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 0 | 4
  White | 12 | 8 | 3 | 23
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 1 | 8
Region of Enrollment [Number; unit: participants]
  United States | 18 | 16 | 4 | 38
Estrogen Receptor (ER) Type [Count of Participants; unit: Participants]
  ER Positive (ER+) | 18 | 16 | 0 | 34
  ER Negative (ER-) | 0 | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Objective response rate (ORR) will be defined as the proportion of participants whose status is stable disease (SD) or better (complete response (CR), partial response (PR)) at 24 weeks' follow-up as measured by Response Evaluation Criteria in Solid Tumors (RECIST). The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The patient's best response assignment will depend on the achievement of both measurement and confirmation criteria.
Time Frame: Up to 24 weeks
Population: Participants in Group C were off treatment prior to assessment and not included in this analysis
Measure: Number; unit: percentage of participants
Groups:
- Pembrolizumab: Group B: Estrogen Receptor Positive (ER+) participants
  Tamoxifen: 20 mg daily orally (starting at Cycle 1) Vorinostat: 400 mg 5 days every 7 orally (starting at Cycle 1)
  Group B Pembrolizumab: 200 mg every 3 weeks intravenously (starting at Cycle 2)
Arm/Group | Pembrolizumab Group A | Pembrolizumab: Group B | Pembrolizumab Group C
Number analyzed (Participants) | 15 | 13 | 0
percentage of participants | 6.67 | 0 |

2. Primary Outcome: Number of Participants With Treatment-related Adverse Events (AE)
Description: Each patient who received at least 1 dose of any of the study drugs will be assessed periodically for the development of any grade 3 and higher treatment-related toxicity according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4. The investigators will also pay particular attention to pembrolizumab adverse events of clinical interest (ECI), which will predominantly be of immune origin.
Time Frame: Up to 1 year post treatment, approximately 24 months
Measure: Count of Participants; unit: Participants
Groups:
- Pembrolizumab Group B: Estrogen Receptor Positive (ER+) participants
  Tamoxifen: 20 mg daily orally (starting at Cycle 1) Vorinostat: 400 mg 5 days every 7 orally (starting at Cycle 1)
  Group A Pembrolizumab: 200 mg every 3 weeks intravenously (starting at Cycle 2)
Arm/Group | Pembrolizumab Group A | Pembrolizumab Group B | Pembrolizumab Group C
Number analyzed (Participants) | 18 | 16 | 4
Participants
  Anorexia | 0 | 1 | 0
  Fatigue | 1 | 1 | 0
  Thrombocytopenia | 1 | 1 | 1
  Elevated Transaminitis (Liver Enzymes) | 2 | 0 | 0
  Hyponatremia | 1 | 1 | 0
  Stroke | 1 | 0 | 0

3. Secondary Outcome: Duration of Response
Description: The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
Time Frame: Up to 24 months
Population: No participants from Group C achieved an objective response
Measure: Median (Full Range); unit: months
Arm/Group | Pembrolizumab Group A | Pembrolizumab Group B | Pembrolizumab Group C
Number analyzed (Participants) | 15 | 13 | 0
months | 17.0 [6.5 to 21.7] | 8.8 [8.7 to 8.8] |

4. Secondary Outcome: Progression Free Survival
Description: Progression-free survival (PFS) is defined as the length of time during and after the treatment that the participant has achieved an objective response, but does not progress as measured by RECIST v.1.1
Time Frame: Up to 36 months
Population: No participants from Group C achieved an objective response
Measure: Median (Full Range); unit: months
Arm/Group | Pembrolizumab Group A | Pembrolizumab Group B | Pembrolizumab Group C
Number analyzed (Participants) | 15 | 13 | 0
months | 2.57 [1.1 to 21.7] | 2.63 [1.0 to 8.6] |

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the length of time from the start of treatment for participants until death or the study has ended, whichever comes first.
Time Frame: Up to 36 months
Measure: Median (Full Range); unit: months
Arm/Group | Pembrolizumab Group A | Pembrolizumab Group B | Pembrolizumab Group C
Number analyzed (Participants) | 15 | 13 | 4
months | 14.3 [1.0 to 34.8] | 15.0 [3.3 to 34.8] | 7.8 [3.8 to 29.5]

6. Secondary Outcome: Number of Participants With Tumor Responses Calculated by Immune Related Response-Criteria (irRC)
Description: In the irRC, an immune-related Complete Response (irCR) is defined as the disappearance of all lesions, measured or unmeasured, and no new lesions; an immune-related Partial Response (irPR) is defined as a 50% drop in tumour burden from baseline, and immune-related Progressive Disease (irPD) is a 25% increase in tumour burden from the lowest level recorded. All other responses are considered immune-related Stable Disease (irSD). The number of participants with a tumor response of either irCR or irPR will be reported.
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab Group A | Pembrolizumab Group B | Pembrolizumab Group C
Number analyzed (Participants) | 15 | 13 | 4
Participants | 1 | 0 | 0

7. Secondary Outcome: Number of Participants With a Clinical Response (Clinical Benefit) Based on PD-L1 Expression to Epigenetic Immune Priming
Description: PD-L1 protein expression on tumor tissue from pre-treatment and post-Cycle-3 biopsies, and any other tumor biospecimens obtained, were evaluated immunohistochemically. Patients were categorized based on detectable PD-L1 expression as Positive or Negative for expression. Participants with positive PD-L1 expression were then reviewed to determine if a clinical benefit was obtained at cycle 6. Clinical benefit was defined as a complete response or partial response per RECIST 1.1.
Time Frame: Up to 18 weeks, at Cycle 6
Population: All necessary data required for inclusion in this analysis could not be obtained for participants in Group C
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab Group A | Pembrolizumab Group B | Pembrolizumab Group C
Number analyzed (Participants) | 15 | 13 | 0
Participants
  PD-L1 Negative | 14 | 12 |
  PD-L1 Positive | 1 | 1 |
  PD-L1 Positive with clinical benefit at cycle 6 | 0 | 0 |

ADVERSE EVENTS:
Time Frame: Up to 24 months
Groups:
- Pembrolizumab Group A: Estrogen Receptor Positive participants (ER+)
  Tamoxifen: 20 mg daily orally (starting at Cycle 1) Vorinostat: 400 mg 5 days every 7 orally (starting at Cycle 1) Group A: Pembrolizumab: 200 mg every 3 weeks intravenously (starting at Cycle 1)
- Pembrolizumab Group B: Estrogen Receptor Positive participants (ER+)
  Tamoxifen: 20 mg daily orally (starting at Cycle 1) Vorinostat: 400 mg 5 days every 7 orally (starting at Cycle 1) Group B: Pembrolizumab: 200 mg every 3 weeks intravenously (starting at Cycle 2)
- Pembrolizumab Group C: Estrogen Receptor Negative participants (ER-)
  Vorinostat: 400 mg 5 days every 7 orally (starting at Cycle 1) Pembrolizumab: 200 mg every 3 weeks intravenously (starting at Cycle 1)
Arm/Group | Pembrolizumab Group A | Pembrolizumab Group B | Pembrolizumab Group C
All-Cause Mortality (participants affected / at risk) | 1/18 | 0/16 | 0/4
Serious Adverse Events (participants affected / at risk) | 6/18 | 4/16 | 0/4
Other Adverse Events (participants affected / at risk) | 17/18 | 15/16 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab Group A (N=18) | Pembrolizumab Group B (N=16) | Pembrolizumab Group C (N=4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Weight Loss (Investigations) | 0 (0) | 1 (1) | 0 (0)
Acute renal failure (ARF) (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab Group A (N=18) | Pembrolizumab Group B (N=16) | Pembrolizumab Group C (N=4)
Diarrhea (Gastrointestinal disorders) | 6 (16) | 4 (4) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (8) | 4 (10) | 2 (2)
Vomiting (Gastrointestinal disorders) | 6 (6) | 3 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (6) | 4 (5) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0)
Fatigue (General disorders) | 11 (20) | 5 (7) | 4 (8)
Pain (General disorders) | 4 (6) | 2 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 5 (10) | 6 (6) | 4 (5)
Platelet count decreased (Investigations) | 4 (7) | 3 (9) | 1 (4)
Weight loss (Investigations) | 3 (4) | 4 (6) | 2 (3)
Creatinine increased (Investigations) | 2 (2) | 4 (8) | 0 (0)
Dysgeusia (Nervous system disorders) | 4 (8) | 2 (4) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 1 (3) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (3) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 2 (2)
Hot Flashes (Vascular disorders) | 4 (4) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Stomach Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0) | 2 (2)
Edema limbs (General disorders) | 2 (2) | 1 (1) | 0 (0)
Breast Pain (Reproductive system and breast disorders) | 3 (3) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 2 (3)
Hypokalemia (Investigations) | 3 (4) | 2 (2) | 0 (0)
Hyponatremia (Investigations) | 1 (2) | 1 (2) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 0 (0)
Fever (General disorders) | 2 (2) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Hypophosphatemia (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Investigations) | 1 (1) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 1 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was closed early due to insufficient efficacy in an unselected patient population and slow accrual which resulted in small sample sizes by arm. Approximately 29 participants were needed, per arm, for sufficiently powered statistical analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/27/NCT02395627/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-07-28): https://cdn.clinicaltrials.gov/large-docs/27/NCT02395627/Prot_SAP_001.pdf